CLINICAL TRIAL: NCT02162316
Title: A Multicenter, Randomized, Double-blind Comparative Study to Evaluate the Efficacy Between Helicobacter Pylori Eradication Therapy and Motilitone in Functional Dyspepsia
Brief Title: A Study to Evaluate the Efficacy Between Helicobacter Pylori Eradication Therapy and Motilitone in Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Jae Gyu Kim, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HyFu
Record Dates: First submitted 2014-06-11; First posted 2014-06-12 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H.Pylori eradication therapy (Active Comparator): A-cillin®, Pantoline® and Clari® is administered with a tablet of placebo (Motilitone®)
  Interventions: Drug: A-Cilin®, Clari® and Pantoline®
- Motilitone® (Experimental): 30 mg is administered with 3 tablets of placebo (Patoline®, Clari® and A-cilin)
  Interventions: Drug: Motilitone®

INTERVENTIONS:
Drug: Motilitone®
  Arms: Motilitone®
Drug: A-Cilin®, Clari® and Pantoline®
  Arms: H.Pylori eradication therapy

SUMMARY:
This is a clinical study to evaluate the efficacy between Helicobacter pylori Eradication therapy and Motilitone in Functional Dyspepsia

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind comparative clinical study to evaluate the efficacy between Helicobacter pylori Eradication therapy and Motilitone in Functional Dyspepsia

ELIGIBILITY:
Inclusion Criteria:

* Roman III criteria
* One or more conditions are applied: epigastric pain, epigastric burning, bothersome, postprandial fullness or early satiety
* No organic lesion
* Helicobacter pylori infection

Exclusion Criteria:

* has taken prokinetics, H2 antagonists, PPIs, NSAIDs, anticholinergics, antibiotics, antidepressants, anticoagulants within a month
* had a surgery that might affect gastrointestinal motility

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Volunteer global assessment of improvement rate of functional dyspepsia by using 5-Likert scale | 12 weeks
  5-Likert scale
  1. deteriorated
  2. not changed
  3. moderately improved
  4. markedly improved
  5. symptom-free

SECONDARY OUTCOMES:
Volunteer global assessment by using 5-Likert scale | 6 weeks
The improvement rate of 4 types of dyspepsia symptoms | 12 weeks
The change of each score and total score of dyspeptic symptoms | 6, 12 weeks
Assessment of NDI-K Quality of Life | 6,12 weeks
The proportion of the patients who answered "yes for the question about symptom improvement | 6, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Hong, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital; Gwang Ha Kim, M.D., Ph.D., Principal Investigator — Busan National University Hospital; Sang Gyun Kim, M.D., Ph.D, Principal Investigator — Seoul National University Hospital; Hyun Soo Kim, M.D., Ph.D, Principal Investigator — Chonnam National University Hospital; Seong-Woo Jeon, M.D., Ph.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea